CLINICAL TRIAL: NCT05689879
Title: Evaluation of TNF-alpha Antagonists (Infliximab) Withdrawal in Sarcoidosis : a Prospective, Randomized, Controlled Trial
Brief Title: Evaluation of TNF-alpha Antagonists (Infliximab) Withdrawal in Sarcoidosis
Acronym: TAWIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160922
Record Dates: First submitted 2022-05-02; First posted 2023-01-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-04

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Intervention Model Description: Infliximab stop Methotrexate (without exceed 25mg/kg/week) or azathioprine
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMAIN arm (No Intervention): Infliximab 3 to 5 mg/kg every 4-8 weeks, methotrexate 7.5-10 mg/week (or azathioprine 1 mg/Kg/day), steroids < or = 10 mg/day
- STOP arm (Other): Methotrexate 0.3 mg/kg/week (or azathioprine 2 mg/kg/day (or 1 mg/kg/day if intermediary metabolism TMPT) (the dose of methotrexate will not exceed 25mg/kg/week wathever the weight of the patient), steroids < or = 10 mg/d
  Interventions: Drug: STOP arm

INTERVENTIONS:
Drug: STOP arm — TNF-alpha antagonists withdrawal
  Other Names: TNF-alpha antagonists withdrawal
  Arms: STOP arm

SUMMARY:
In severe refractory sarcoidosis not responding to conventional immunosuppressive treatment, the third-line tumor necrosis factor (TNF)-alpha inhibitor infliximab is an alternative. Treatment duration is not known, although it has been suggested that relapse rates after withdrawal could be high. We hypothesize that a prolonged course of TNF-alpha would be better for maintaining remission in sarcoidosis.

The population consists of histologically-proven adults sarcoidosis patients who were treated with infliximab and are in remission for at least 6 months with less than or equal to 10 milligrams of steroids (prednisone).

The present study is a phase 3, prospective, randomized, parallel groups, comparative, open-labelled 2 arms study superiority trial comparing a STOP to a REMAIN strategy. Patients will be randomized in the 2 groups in a 1:1 ratio.

DETAILED DESCRIPTION:
The screening visit takes place between 60 days and until the baseline visit. The investigator will first check that the patient meets the inclusion criteria and does not present exclusion criteria. Before enrolment and randomization, all patients will receive comprehensive information and provide written consent.

Visit schedule:

* Baseline visit
* Follow-up Visits In the REMAIN arm: visits will be performed each 4-8 weeks depending on the infliximab interval. In the STOP arm, visits will be performed every 8 weeks, and in case of relapse (until M12+/- 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age superior or equal to 18 years
* Clinical and radiological presentation consistent with sarcoidosis
* Presence of non-caseating granulomas in at least one organ
* Exclusion or other causes of granulomas
* Infliximab treatment for at least 6 months
* Steroid dosage < or equal to 10 mg/day for at least 6 months
* No activity of the disease (ePOST score 0) for at least 6 months
* Normal ACE (angiotensin converting enzyme) and serum calcemia level
* Signed informed consent
* Affiliated to the National French social security system
* As infliximab is the most used TNF-alpha antagonists, we decided to include only patients treated with infliximab to increase the homogeneity.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Positive IGRA (Interferon Gamma Release Assays) test without previous antituberculous antibiotherapy
* Active infection
* Patients with moderate to severe heart failure (NYHA class III/ IV)
* Severe liver function disorders
* Alcoholism
* Severe kidney function disorders
* Pre-existing blood dyscrasias
* History of cancer in the 5 years before enrolment (except for cutaneous non melanoma cancers)
* Concurrent vaccination with live vaccines during therapy
* Inability to understand information about protocol
* Adult subject under legal protection or unable ton consent
* Absence of effective contraceptive method for men and women for duration of the study and 6 months after the end of participation
* Concomitant participation to another biomedical research (only Category 1 trial according to the french law)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To compare 2 strategies of remission maintenance in patients who are in remission after infliximab administration | 12 months
  Percentage of patients with major relapse (reappearance or worsening of the disease with a ePOST score >0 and involvement of at least one major organ, a life-threatening situation, or both or relapse non responsive to mild treatment intensification) between enrolment and month 12.
  Major organs are nervous system, heart, kidneys, muscles and lungs. Mild treatment intensification is defined by increasing the dosage of steroids at more than 20 milligrams/day.
  The primary criterion will be assessed at each visit, in case of relapse and at the end of follow-up (M12).

SECONDARY OUTCOMES:
To compare the percentage of patients with minor relapses in the 2 groups | 12 months
  Percentage of patients with minor relapse (reappearance or worsening of the disease with a ePOST score > 0 not corresponding to the definition of major relapse) at months 12.
To compare the rates of adverse events | 12 months
  All adverse events occurred between enrolment and Month 12, will be noted with special attention to infection, haematological toxicities and cancers.
To determine which are the predictors of relapses | 12 months
  Percentage of patients with a previous heart involvement at inclusion
To determine which are the predictives of relapses | 12 months
  Percentage of patients with nervous system involvement at inclusion
To determine which are the relapsing predictors | 12 months
  Percentage of patients with hypermetabolism elsewhere consistent with sarcoidosis localization in positron emission tomography scan (PET scan) at inclusion
To determine which are the prediction of relapses | 12 months
  Serum ACE (angiotensin converting enzyme) level at inclusion
To compare results of Short Form (36) Health Survey in the 2 groups | 12 mois
  Quality of life will be assessed by SF-36 (Short Form (36) Health Survey) at inclusion, Month 6 and Month 12 (score from 0 to 100, the higher score is the better).
Compare results of Nottingham scale of each groups | 12 mois
  Quality of life will be assessed by Nottingham scale at inclusion, Month 6 and Month 12 (score from 0 to 38, the higher score is the worse) .
To compare results of Fatigue Assessment Scale in the 2 groups | 12 mois
  Quality of life will be assessed by Fatigue Assessment Scale (FAS, Patel 2000) at inclusion, Month 6 and Month 12 (score from 10 to 50, the higher score is the worse) .

CONTACTS AND LOCATIONS:
Overall Officials: Fleur COHEN AUBART, PHD, Study Director — Internal Medicine Department 2 - Hôpital Pitié-Salpêtrière
Locations (1):
- Hôpital de la Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No